CLINICAL TRIAL: NCT00011908
Title: A Phase I Clinical Trial of Immunotherapy With Humanized LL2 IgG (Epratuzumab) in Patients With Systemic Lupus Erythematosus
Brief Title: Humanized LL2IGG to Treat Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 010108; 01-AR-0108
Record Dates: First submitted 2001-03-03; First posted 2001-03-05 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Safety; B-Lymphocyte Depletion; Anti-CD22; Response; Efficacy; Lupus; Immunotherapy
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — epratuzumab

INTERVENTIONS:
Drug: hLL2 (Epratuzumab)

SUMMARY:
This study will examine the safety of a new genetically engineered antibody called hLL2 (epratuzumab) in patients with systemic lupus erythematosus (SLE). It will also evaluate whether hLL2 can lessen overall disease activity in SLE or kidney damage in patients with lupus nephritis.

Patients 18 years of age and older with mild to moderately active SLE may be eligible for this study. Candidates will be screened with blood and urine tests, a chest X-ray, electrocardiogram (EKG), tuberculin skin test, and screening tests for certain cancers.

All participants will receive weekly infusions of hLL2 for 4 weeks. The drug is given through a catheter (small plastic tube) placed through a needle in an arm vein. Each infusion takes about 2 hours, after which the patient is observed in the clinic for 1 to 2 hours before being discharged from the clinic.

The first 3 patients in the study will receive the lowest of three different doses used in the study. If this dose is well tolerated, the next 5 patients will receive a higher dose. If the second dose is tolerated, the last 5 patients will be given the highest dose. If any serious problems are encountered at a dose, patients in the next group will receive either the same or lower dose before being advanced to the next level. Patients in the first group will continue taking prednisone at their regular dose. All other patients will have their prednisone tapered gradually, if their condition permits. Patients who have a disease flare may have their prednisone increased for up to 2 weeks, followed by a gradual taper. If the flare is severe or does not respond to the increased prednisone, the patient will be taken off the study and treated to control the disease.

Patients will be evaluated at various intervals for up to 8 weeks after the last dose. Several of the screening tests will be repeated throughout the study. No more than 500 ml of blood-the equivalent of a single blood donation-will be collected during a 2-month period. Participants may also be asked to undergo the following optional procedures before starting treatment, 1 week after the last dose and 8 weeks after the last treatment dose:

* Bone marrow aspiration - to collect cells from the bone marrow. The hip area is anesthetized and a special needle is used to draw bone marrow from the hipbone.
* Tonsil biopsy - The area to be biopsied is numbed with a local anesthetic and small pieces of tissue will be removed with a special type of forceps. (The procedure may be done under general anesthetic.)
* Magnetic resonance imaging (MRI) of the abdomen - The patient lies on a table within a metal cylinder (the MRI scanner) for about 30 to 40 minutes while images are obtained with the use of a strong magnetic field and radio waves.

DETAILED DESCRIPTION:
This is a pilot study to evaluate the safety and tolerance of hLL2 (epratuzumab), a humanized anti-CD22 monoclonal antibody, in patients with systemic lupus erythematosus (SLE).

B-lymphocytes play a major role in initiating and maintaining the underlying immunopathological mechanisms of SLE. In addition to producing autoantibodies, they also serve as antigen presenting cells and are able to disrupt peripheral T lymphocyte tolerance. Furthermore, B lymphocyte depletion ameliorates disease activity in animal models of SLE. Therefore, targeted depletion of B-lymphocytes may be of therapeutic benefit in human SLE.

hLL2 (epratuzumab) is a humanized monoclonal antibody that binds to CD22, a surface antigen expressed exclusively on B-lymphocytes. Clinical studies in patients with B cell lymphomas have shown that epratuzumab is safe and well tolerated across a wide range of doses. Although the exact mechanism is unknown, indirect evidence suggests that the antibody is depleting target B lymphocytes. Epratuzumab is made available by Immunomedics, Inc., and will be used under an investigator (NIH)-initiated IND.

In this open-label, Phase I study, up to 20 patients with moderately active SLE may be enrolled. Patients will be treated with weekly infusions of hLL2 in one of three different dosing groups [(240 mg/m(2), 360 mg/m(2), 480 mg/m(2)] for 4 weeks, and followed for 8 weeks after the last dose.

The primary objective is to determine the safety and tolerability of hLL2 in patients with SLE. In addition to safety data, clinical and laboratory data will also be collected for preliminary evaluation of the effectiveness of hLL2 in SLE and to assess the effect of hLL2 on B and T lymphocytes in the lymphoid organs and the peripheral blood. If the treatment is safe and there is preliminary evidence of efficacy, this regimen could be used in controlled trials in the future.

ELIGIBILITY:
INCLUSION/EXCLUSION CRITERIA

Patients must be at least 18 years of age at entry.

Patients must give written informed consent prior to entry in the protocol.

Patients must fulfill at least 4 criteria for SLE as defined by the American College of Rheumatology.

Patients with active lupus not requiring immediate immunosuppressive therapy other than oral prednisone less than or equal to 0.3 mg/kg/day (or its equivalent) are eligible. Active lupus is defined by any of these three (a-c) sets of criteria:

a. Chronic proliferative glomerulonephritis with partial or no response to at least 6 months of adequate immunosuppressive therapy (with pulse methylprednisolone, cyclophosphamide, azathioprine, cyclosporine, mycophenolate mofetil or high dose daily corticosteriods), and

i. less than 50% increase in creatinine compared from lowest level during treatment

ii. proteinuria less than or equal to 1.5 times the baseline before treatment

iii less than or equal to 2+ cellular casts in the urinary sediment (on a scale of 0-4),

b. Newly diagnosed proliferative glomerulonephritis with

i. a biopsy showing crescents and/or necrosis in less than 25% of the glomeruli and minimal or no interstitial fibrosis

ii. proteinuria less than or equal to 3.5 gm/day and albumin greater than or equal to 3.0 gm/dL

iii. creatinine less than or equal to 1.5 mg/dL,

c. Patients with moderately active extra-renal lupus defined as a SLEDAI score between 3-10.

Patients who have renal and extrarenal disease will be included in the study if they fulfill any of the above inclusion criteria. Their SLEDAI score will be determined based on the extrarenal features of their disease (non-renal SLEDAI).

Patients must have serum dsDNA level greater than 2 times the upper limit of normal or IgG anticardiolipin antibody levels greater than or equal to 20 GPL.

Patients must have stable doses of prednisone less than or equal to 0.3 mg/kg/day (or its equivalent) for at least 2 weeks before the first treatment.

Pregnant or lactating women are not eligible.

Women of childbearing potential and fertile men who are not practicing or who are unwilling to practice birth control during and for a period of three months after the completion of the study are excluded from the study.

Patients who have had any therapy with human or murine antibodies or any experimental therapy within 3 months are not eligible.

Patients who have had therapy with cyclophosphamide, pulse methylprednisolone or IVIg within 4 weeks or azathioprine, mycophenolate mofetil, cyclosporine or methotrexate within 2 weeks of first study treatment are not eligible.

Patients who have an initiation or a change in the dose of an ACE-inhibitor within 2 weeks of first study treatment are not eligible.

Patients must not have an allergy to murine or human antibodies.

Patients with serum creatinine greater than 2.5 mg/dL are excluded.

Patients with 24 hour proteinuria greater than 5.5 gm/day are excluded.

Patients who have active severe CNS lupus (encephalopathy, cerebrovascular accident, transverse myelitis, severe depression, psychosis) are not eligible.

Patient who have a history of thrombosis or recurrent 2nd trimester abortions (3 or more) and elevated levels of anti-cardiolipin antibodies or lupus anticoagulant unless the patient is on anticoagulation are not eligible.

Patients who have a history of malignancy with the exception of basal cell carcinoma of the skin are not eligible.

Patients who have a serious active infection are not eligible.

Patients who have active hepatitis B, hepatitis C or HIV infection are not eligible.

Patients who have a CD4+ lymphocyte count less than 200 are not eligible.

Patients with WBC less than 2000 or ANC less than 1500 or Hgb less than 8.0 or platelets less than 50,000/microliters or transaminases greater than 2 times the upper limit of normal or alkaline phosphatase greater than 2 times the upper limit of normal are not eligible.

Patients must not have a significant concurrent medical condition that, in the opinion of the principal investigator, could affect the patient's ability to tolerate or complete the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2001-02; Study Completion 2003-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Velasquez WS, Cabanillas F, Salvador P, McLaughlin P, Fridrik M, Tucker S, Jagannath S, Hagemeister FB, Redman JR, Swan F, et al. Effective salvage therapy for lymphoma with cisplatin in combination with high-dose Ara-C and dexamethasone (DHAP). Blood. 1988 Jan;71(1):117-22. PMID 3334893
- [Background] Klimo P, Connors JM. Updated clinical experience with MACOP-B. Semin Hematol. 1987 Apr;24(2 Suppl 1):26-34. PMID 2438779
- [Background] Dana BW, Dahlberg S, Miller TP, Hartsock RJ, Balcerzak S, Coltman CA, Carden JO, Hartley K, Fisher RI. m-BACOD treatment for intermediate- and high-grade malignant lymphomas: a Southwest Oncology Group phase II trial. J Clin Oncol. 1990 Jul;8(7):1155-62. doi: 10.1200/JCO.1990.8.7.1155. PMID 1694233